CLINICAL TRIAL: NCT07364916
Title: Effect of Water Flossing on Gingival Inflammation Around Single Implants: Randomized Clinical Trial
Brief Title: Effect of Water Flossing on Gingival Inflammation Around Single Implants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Amal Jamjoom, BDS, MS., Assistant Professor at KAU, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 129-11-24
Record Dates: First submitted 2025-12-13; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Peri Implant Mucositis
Keywords: Peri- implant; Mucositis; Water irrigation; Water flosser
MeSH Terms: conditions — Mucositis | interventions — Toothbrushing

STUDY DESIGN:
Intervention Model Description: Two groups of implant patients will be randomly allocated to one of 2 interventions; one group will brush only. The other group will brush and use the water flosser around the implant with mucositis.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water flosser (Experimental): The use of a water flosser+ brushing around implants with mucositis
  Interventions: Device: Water flosser
- Control (Active Comparator): Brushing and using the string floss.
  Interventions: Device: Tooth brush and string floss

INTERVENTIONS:
Device: Water flosser — Water irrigation device
  Arms: Water flosser
Device: Tooth brush and string floss — The control group will use the toothbrush and the regular string floss.
  Arms: Control

SUMMARY:
This study aims to evaluate the effect of water floss in reversing peri- implant mucositis around dental implants

DETAILED DESCRIPTION:
Patients will be assigned for two clinical appointments, the first visit is for baseline charting, probing depth will be recorded on six sites per implant, using a standardized periodontal probe and the presence or absence of bleeding will be recorded. Disclosing tablets will be utilized to

Confirm the presence or absence of plaque around teeth and the implant. Patients (Group A) will be given a water floss, with verbal and written instructions to use the water floss, twice daily for 2 minutes, along with brushing, while Group B will be instructed to brush with a manual brush alone, twice daily for 2 minutes. After two weeks, in the second visit, the implant site is re-evaluated to monitor the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Medically cleared
* Have at least one implant-supported crown.

Exclusion Criteria:

1. Smoking
2. Any systemic or localized illness that would interfere with dental implant therapy
3. On medications
4. Pregnancy
5. History of periodontitis/ or peri-implant disease
6. Poor oral hygiene
7. Probing depth is >5

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Bleeding on Probing | 2 and 4 weeks
  The disappearance of bleeding upon probing with the University of North Carolina-15 mm (UNC-15) periodontal probe. It is done at the same time as probing the pocket depths. It is done at six sites per implant-presence of bleeding = 1, absence = 0 -at each site.
Plaque Index of Silness and Loe | 4 weeks
  Score Description 0 No plaque 1 A thin film of plaque adhering to the free gingival margin and adjacent area of the implant; not visible to the naked eye but detectable by probe 2 Moderate accumulation of soft deposits visible to the naked eye within the gingival pocket and/or on the implant and gingival margin | 3 Abundant soft matter within the gingival pocket and/or on the implant and gingival margin |

SECONDARY OUTCOMES:
Probing Pocket Depths (PPD) | 4 weeks
  The PPD will be recorded at baseline visit using the UNC-15 periodontal probe, at 2 weeks, and at 4 weeks. Pocket depths around implants should usually be around 1-4 mm. Pockets that are deeper than 4 mm or are 4 mm or less but with bleeding will be recorded as abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: Amal G Jamjoom, Principal Investigator — King Abdulaziz University

IPD SHARING:
Plan to Share IPD: Yes
Access to de-identified individual participant data will be granted to qualified researchers who submit a scientifically sound proposal outlining the research objectives and planned analyses. Requests will be reviewed by the principal investigator to ensure alignment with the original study aims, ethical approval, and data protection requirements. Approved applicants will be required to sign a data use agreement prior to data release. Data will be provided in a secure, de-identified format and used solely for the approved purpose.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD will be available beginning 6 months after publication of the primary results and will remain available for up to 5 years thereafter.
Access Criteria: Requests for access to the IPD should be directed to the corresponding author. Data will be shared in a secure format following approval of the request and execution of a data use agreement.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2026-01-18): https://cdn.clinicaltrials.gov/large-docs/16/NCT07364916/Prot_SAP_000.pdf